CLINICAL TRIAL: NCT04726592
Title: Randomized Double Blinded Monocentric Study Evaluating the Efficacy of CLORazepate for the Treatment of MIGraine Attack in the Emergency Room
Brief Title: Efficacy of CLORazepate for the Treatment of MIGraine Attack in the Emergency Room
Acronym: CLORMIG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: It has been determined that continuing with enrollments in this study is no longer justified due to the lack of significant impact on the expected outcomes.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P170903J
Record Dates: First submitted 2021-01-24; First posted 2021-01-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-10

CONDITIONS: Migraine; Migraine Without Aura; Migraine With Aura; Headache
MeSH Terms: conditions — Migraine Disorders; Migraine without Aura; Migraine with Aura; Headache | interventions — Clorazepate Dipotassium; Ketoprofen; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Placebo Comparator): placebo and standard care :
  * Placebo IV
  * Ketoprofen 100 mg IV (if nausea-vomiting)
  * Metoclopramide 10 mg IV(if nausea-vomiting)
  Interventions: Drug: Placebo; Drug: Ketoprofen; Drug: Metoclopramide
- Experimental arm (Experimental): clorazepate and standard care :
  * Clorazepate 20 mg IV
  * Ketoprofen 100 mg IV (if nausea-vomiting)
  * Metoclopramide 10 mg IV(if nausea-vomiting)
  Interventions: Drug: Clorazepate Dipotassium; Drug: Ketoprofen; Drug: Metoclopramide

INTERVENTIONS:
Drug: Clorazepate Dipotassium — Clorazepate Dipotassium : 20 mg intravenous injection
  Other Names: TRANXENE
  Arms: Experimental arm
Drug: Placebo — Placebo IV
  Arms: Control arm
Drug: Ketoprofen — Ketoprofen 100 mg IV
Drug: Metoclopramide — Metoclopramide 10 mg IV

SUMMARY:
The purpose of this study is to evaluate the efficacy of clorazepate in addition to the usual medication for treating migraine attack in the emergency room

DETAILED DESCRIPTION:
Each patient will receive the usual migraine treatment: IV ketoprofen 100 mg and, if he suffers nausea and/or vomiting, additional IV metoclopramide 10 mg.

Depending on randomization assignment, patient will receive additional placebo (standard treatment arm) or additional IV Clorazepate 20 mg (study arm). The central pharmacy will be responsible for preparing the medications, using a double-blind protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70
* Patient suffering migraine or probable migraine (diagnosis made by neurologist according to IHCD3)
* Present migraine attack lasting ≤ 72 hours
* Headache intensity moderate or severe on the verbal ordinal scale (4 levels: no headache, mild, moderate or severe)
* Patient requiring parenteral treatment
* Affiliation to the French Health-care System "sécurité sociale"

Exclusion Criteria:

* abnormalities of neurological exam, seizure, fever (≥ 38°C), and/or SBP≥180 and/or DBP≥110 mmHg
* suspicion of secondary headache
* inability to understand the consent or scales
* pregnancy or breast-feeding
* known respiratory or liver insufficiency
* acute alcohol consumption or alcoholism
* myasthenia
* Patient requiering treatment with sumatriptan SC, particularly in the event of failure of an anti-inflammatory drug at an effective dose taken within 6 hours
* recent use of benzodiazepines (< 24h diazepam, clonazepam, clorazepate ; < 6h alprazolam, lorazepam, midazolam)
* recent use of pain killers (< 2h)
* contraindication to any of the investigational medication
* contraindication to intravenous access
* previous participation to this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Pain relief | 2 hours
  Percentage of patients "pain-relief" 2 hours after administration of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lariboisière, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No